CLINICAL TRIAL: NCT00200187
Title: A Randomized Study of the Efficacy of Low Venous Pressure General Anesthesia Versus Combined Spinal-Epidural Anesthesia in Decreasing Blood Loss During Radical Retropubic Prostatectomy
Brief Title: A Randomized Study of the Efficacy of Low Venous Pressure General Anesthesia Versus Combined Spinal-Epidural Anesthesia in Decreasing Blood Loss During Prostate Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-003
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Prostate Cancer
Keywords: Prostatectomy; Anesthesia; Blood Loss
MeSH Terms: conditions — Prostatic Neoplasms; Hemorrhage

INTERVENTIONS:
Procedure: low venous pressure general anesthesia
Procedure: combined spinal-epidural anesthesia

SUMMARY:
You are being asked to join the study because you have early stage prostate cancer and will have your prostate removed. The purpose of this study is to compare blood loss during surgery among two types of anesthesia. One type is general anesthesia. It puts you in a deep enough sleep that you will not feel anything. It also keeps your blood pressure low, which might decrease bleeding. The second type is combined spinal-epidural anesthesia. For this type, a small catheter is placed in your spinal canal through your back. Anesthesia given through the catheter makes your body numb from the waist down, so the sleep you would be in is not so deep. Your blood pressure would remain in your normal range. After surgery, the catheter remains in place to treat your pain, but your body would not be numb. When you wake up after general anesthesia, you would receive pain medicine through a vein in your arm.

Both types are used at Memorial Hospital. They are accepted forms of anesthesia. We will be looking at blood loss between these two types for patients having their prostate removed. We also want to learn about the side effects of each anesthesia type, and assess pain that you experience after surgery.

DETAILED DESCRIPTION:
This is a prospective randomized trial comparing the efficacy of a low venous pressure general anesthesia (LVPGA) technique vs. combined spinal-epidural anesthesia (CSE) in decreasing intraoperative blood loss in patients undergoing open radical retropubic prostatectomy (RRP) for newly diagnosed clinically localized adenocarcinoma of the prostate. The study design involves the enrollment of 246 patients scheduled for RRP. To control for surgeon technique in the varibility of intraoperative blood loss, the study will be limited to the patient population of two surgeons who perform greater than 150 radical prostatectomies per year. Patients will be stratified for each surgeon and will be randomized to receive either a LVPGA or CSE. Preoperatively patients will be encouraged to donate autologous blood as is the current practice at MSKCC. Perioperative measurement and management of fluid administration, estimation of blood loss and urine output, and transfusion criteria will be standardized for both anesthesia groups. Transfusion of blood products will be at the discretion of the attending surgeon and anesthesiologist following the guidelines described in the protocol. Autologous blood will not routinely be transfused back if the hemoglobin is >= 8.0 and the patient is not symptomatic. Patients randomized to the CSE arm will also receive postoperative epidural analgesia, while patients randomized to LVPGA will receive intravenous PCA analgesia as per our current standard of care. Pain relief will be assessed by a standardized pain scale and recorded in the PACU and then twice daily until discharge. All patients will receive routine preoperative evaluation, as well as routine intraoperative and postoperative monitoring and care. All patients will be placed on a routine postoperative pathway. The MSKCC Morbidity/Mortality DMT Documentation System will be utilized to document postoperative complications as per our routine practice. The Surgical Secondary Events (SSE) program is designed to provide risk adjusted postoperative morbidity and mortality data for institutional comparisons and as a decision support project, generating, reporting and analyzing events to promote change and improvement in patient management. SSE are grouped in 6 grades depending on the severity of the complication and the treatment requirements: Grade 0, no event observed beyond 30 days postop. Grade 1, use of oral medications, bedside interventions to treat an event. Grade 2, use of I.V. medications, TPN, enteral nutrition, or blood transfusion to treat an event. Grade 3, interventional radiology, therapeutic endoscopy, intubation, angiography or operation required to treat an event. Grade 4, residual and lasting disability requiring major rehabilitation or organ resection. Grade 5, event resulting in death of patient.

ELIGIBILITY:
Inclusion Criteria:

* They are scheduled for RRP by Drs. Scardino or Eastham.
* They speak English in order to cooperate during CSE if randomized to such arm.
* They have clinically localized disease, clinical stage < cT3NxM0 (1997 TNM), any Gleason grade
* Must be willing to receive blood products or blood if deemed clinically necessary
* Must be willing to receive epidural or general anesthesia
* All subjects must be age 18 or older
* Patient or the patient's legally acceptable representative must sign and date informed consent PRIOR to any study related procedures being performed.
* Patient must have an MRI of the prostate done at MSKCC prior to RRP.

Exclusion Criteria:

* Prior history of significant cardiac disease (defined as unstable angina, coronary artery stent placement within 8 weeks of surgery, MI within 6 months of surgery, known history of cardiomyopathy, congestive heart failure or significant valvular heart disease), insulin dependent diabetes mellitus, or clinically significant carotid artery disease.
* Presence of renal insufficiency (define by creatinine level > 1.6 mg/dl).
* Prior radiation therapy to the pelvis or prostate
* History of bleeding tendencies, hemorrhagic diathesis, or known primary or secondary hematological disease such as chronic renal failure, Von Willebrand disease, and thrombocytopenia among others.
* History of lumbar spine disease or peripheral neurological conditions that may contraindicate use of CSE anesthesia.
* Prior transurethral resection of the prostate or a suprapubic prostatectomy
* Prior history of an abdominal perineal resection or local excision of a colorectal cancer
* Patients requiring anticoagulation due to a pre-existing medical illness or increased risk for thromboembolic events such as prior history of pulmonary embolus, morbid obesity, atrial fibrillation, mechanical heart valve, etc.
* History of morphine allergy
* History of fentanyl allergy
* History of allergy to local anesthetics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246
Dates: Start 2005-02; Study Completion 2007-01

PRIMARY OUTCOMES:
Aim #1: To determine whether LVPGA reduces blood loss by >= 300 ml versus CSE in patients undergoing open RRP
Aim #2: To compare transfusion rates of autologous and allogenic blood between the two anesthesia groups
Aim #3: To identify differences in pattern of blood loss in the two groups according to different surgical stages
Stage I: Pelvic Lymph node dissection: From skin incision to completion of pelvic node dissection
Stage II: Prostatectomy: From endopelvic fascia opening to completion of prostatic bed hemostasis after the prostate is removed
Stage II a: Dorsal venous complex control: From endopelvic fascia opening to beginning of nerve bundles dissection (or ligature in case they were not preserved)
Stage II b: Nerve bundles dissection and prostate removal: From the beginning of nerve bundles dissection to completion of prostatic bed hemostasis after the prostate is removed
Stage III: Urinary tract reconstruction: From bladder neck reconstruction to completion of skin closure

SECONDARY OUTCOMES:
To compare postoperative complication type, incidence and grade experienced by the two groups. The current MSKCC morbidity and mortality definitions and grading system will be utilized
To compare the efficacy of pain control postoperatively in the two groups (epidural PCA versus intravenous PCA+ NSAID's)
To compare length of hospital stay for the two groups
To prospectively evaluate the relationship of pelvimetry, urethral length and prostatic veins size on MRI 1 to intraoperative blood loss and complications

CONTACTS AND LOCATIONS:
Overall Officials: Sherri M Donat, MD, FACS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://mskcc.org